CLINICAL TRIAL: NCT01115101
Title: A Randomized Controlled Trial: Pain Management After Cesarean Section: Oxycodon vs. Intravenous Piritramide
Brief Title: Superiority Study for Pain Treatment After Cesarean
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Max Dieterich (Other)
Collaborators: University of Rostock (Other)
Responsible Party: Sponsor-Investigator, Max Dieterich, Dr. Max Dieterich, University of Rostock
Organization: University of Rostock (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KJ-2009-MD
Record Dates: First submitted 2010-04-27; First posted 2010-05-04 (Estimated); Results first posted 2013-02-15 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-10

CONDITIONS: Pain
Keywords: pain after cesarean; visual analog scale; oxycodon; piritramid
MeSH Terms: conditions — Pain | interventions — Pirinitramide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxycodon (Experimental)
  Interventions: Drug: Oral Oxycodon
- Patient controlled analgesia (PCA) device with Pritramid (Active Comparator)
  Interventions: Drug: Piritramid

INTERVENTIONS:
Drug: Oral Oxycodon — Patients assigned to the oral analgesia group received 20mg oxycodon at fixed intervals: 2 hours (h) and between 12h and 14h after cesarean.
  Arms: Oxycodon
Drug: Piritramid — Patients assigned to the PCA group received a single use intravenous PCA device (Vygon, Medical Products, Aachen, Germany) with a 30ml deposit of 9% sodium chloride solution containing 60mg piritramide. Bolus injection of 0.5ml was administered by the patient herself if needed, with a lock out interval of 5 minutes
  Patients assigned to the oral analgesia group received 20mg oxycodon at fixed intervals: 2 hours (h) and between 12h and 14h after cesarean. The PCA was discontinued after 24 hours or earlier if demanded.
  Arms: Patient controlled analgesia (PCA) device with Pritramid

SUMMARY:
The purpose of this study is to investigate adequate pain treatment for patients after cesarean. In this study oral opioids were compared to intravenous opioids as they are supposed to provide superior pain control.

DETAILED DESCRIPTION:
Pain management after cesarean is an important topic for women. Pain during and after surgery is their greatest concern.

After surgery quick mobilization is important to take care of the newborn. When using a patient controlled analgesia (PCA) device mobilization is limited and women can not meet their expectations to take care of the newborn. Oral analgesia in comparison offers superior patient satisfaction.

This trial was conducted to investigate the effectiveness of both treatment options and improve patients pain management and overall content after cesarean.

ELIGIBILITY:
Study participation was offered to all pts. aged > 18 years in labor and delivery for elective or unplanned secondary cesarean in the 37th or higher week of gestation.

Inclusion Criteria:

* cesarean in spinal anesthesia,
* no history of opioid or metamizol treatment
* written consent
* ability to use a Patient-controlled analgesia device

Exclusion Criteria:

* cesarean in general anaesthesia
* use of peridural catheter for pre-, peri- or post cesarean analgesia
* additional post cesarean metamizol use
* allergy/hypersensitivity to morphine, oxycodon, acetaminophen or ibuprofen
* chronic use of general anaesthesia
* history of known pain syndrome

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2009-07; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Max Dieterich, MD, Principal Investigator — University of Rostock, Department of Obstetrics and Gynecology
Locations (1):
- University of Rostock, Department of Obstetrics and Gynecology, Rostock, Mecklenburg-Vorpommern, Germany

REFERENCES:
- [Background] Stamer UM, Wiese R, Stuber F, Wulf H, Meuser T. Change in anaesthetic practice for Caesarean section in Germany. Acta Anaesthesiol Scand. 2005 Feb;49(2):170-6. doi: 10.1111/j.1399-6576.2004.00583.x. PMID 15715617
- [Background] Davis KM, Esposito MA, Meyer BA. Oral analgesia compared with intravenous patient-controlled analgesia for pain after cesarean delivery: a randomized controlled trial. Am J Obstet Gynecol. 2006 Apr;194(4):967-71. doi: 10.1016/j.ajog.2006.02.025. PMID 16580284
- [Background] Gammaitoni AR, Galer BS, Bulloch S, Lacouture P, Caruso F, Ma T, Schlagheck T. Randomized, double-blind, placebo-controlled comparison of the analgesic efficacy of oxycodone 10 mg/acetaminophen 325 mg versus controlled-release oxycodone 20 mg in postsurgical pain. J Clin Pharmacol. 2003 Mar;43(3):296-304. doi: 10.1177/0091270003251147. PMID 12638399
- [Background] Carvalho B, Cohen SE, Lipman SS, Fuller A, Mathusamy AD, Macario A. Patient preferences for anesthesia outcomes associated with cesarean delivery. Anesth Analg. 2005 Oct;101(4):1182-1187. doi: 10.1213/01.ane.0000167774.36833.99. PMID 16192541
- [Derived] Dieterich M, Muller-Jordan K, Stubert J, Kundt G, Wagner K, Gerber B. Pain management after cesarean: a randomized controlled trial of oxycodone versus intravenous piritramide. Arch Gynecol Obstet. 2012 Oct;286(4):859-65. doi: 10.1007/s00404-012-2384-5. Epub 2012 May 24. PMID 22622852

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment between July 2009 and November 2009. Of 1112 patients 257 met the inclusion criteria and 239 agreed to participate
Groups:
- Oxycodon: Patients randomized to the oral analgesia group received 20mg oxycodone at fixed intervals at 2 and 12 hours after cesarean section (CS).
- Patient Controlled Device With Pritramid: Patients assigned to the Patient-controlled analgesia (PCA) group received a single use i.v. PCA device (2mg piritramide/ml 0.9% saline, Vygon, Medical Products, Aachen, Germany). A patient initiated i.v. bolus injection contained 1mg piritramide with a lock out interval of 5 minutes. The maximum dose was limited to 30mg piritramide equivalent to 40mg oxycodone total dose.
Period: Overall Study
Arm/Group | Oxycodon | Patient Controlled Device With Pritramid
Started | 113 | 126
Completed | 113 | 126
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Oxycodon: Patients randomized to the oral analgesia group received 20mg oxycodone at fixed intervals at 2 and 12 hours after CS.
- Patient Controlled Device With Pritramid: Patients assigned to the PCA group received a single use i.v. PCA device (2mg piritramide/ml 0.9% saline, Vygon, Medical Products, Aachen, Germany). A patient initiated i.v. bolus injection contained 1mg piritramide with a lock out interval of 5 minutes. The maximum dose was limited to 30mg piritramide equivalent to 40mg oxycodone total dose.
- Total: Total of all reporting groups
Arm/Group | Oxycodon | Patient Controlled Device With Pritramid | Total
Number analyzed (Participants) | 113 | 126 | 239
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 113 | 126 | 239
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.5 (5.9) | 29.8 (5.1) | 29.2 (5.5)
Gender [Count of Participants; unit: Participants]
  Female | 113 | 126 | 239
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 113 | 126 | 239

OUTCOME MEASURES:

1. Primary Outcome: Difference of Pain Scores on the Visual Analog Scale
Description: The primary outcome measure was the change in patients assessment of pain after cesarean (CS) from baseline.
  For pain assessment a visual analog scale (VAS) was used. Women were asked to quantify pain using an eleven point numerical rating score from 0 to 10, with 0 indicating no pain, and 10 the worst pain.
  Single value were calculated (averaged).
Time Frame: Pain level was evaluated before therapy (2h after CS), 12h, 24h, 32h, 40h, 48 and 72h after CS.
Population: The sample size (intention to treat) was computed to detect a difference in VAS score at 24h of 1.2 (30% reduction) at a power of 80%, a two-sided significance level of 0.05.
Measure: Mean (Standard Deviation); unit: VAS score at 24 hours
Arm/Group | Oxycodon | Patient Controlled Device With Pritramid
Number analyzed (Participants) | 113 | 126
VAS score at 24 hours | 5.88 (2.01) | 4.85 (2.23)
Statistical Analysis 1: Comparison: Oxycodon vs Patient Controlled Device With Pritramid; The sample size of n=120 was computed to detect a difference in VAS score at 24h of 1.2 (30% reduction) at a power of 80%, a two-sided significance level of 0.05. Because measurements were made several times on the same patients within in two independent groups, GLM Repeated Measurement procedure was applied to test null hypotheses about the effects of both the between-subject factor (study group) and the within-subject factor (time); Test type: Non-Inferiority or Equivalence — VAS score at 24h were defined as primary endpoint because of the expectation of the maximal effect at this time. Testing for differences of continuous variables between the study groups at baseline was accomplished by the 2-sample t test for independent samples or the Mann-Whitney U test, as appropriate; p < 0.05, Chi-squared; Test selection was based on evaluating the variables for normal distribution employing the Kolmogorov-Smirnov test; Mean Difference (Net) = 0.05, Standard Error of Mean 0.05

2. Secondary Outcome: Subgroups
Description: Secondary Outcome Measures were to identify subgroups in benefit of either therapy.
Time Frame: 6 month
Reporting Status: Not Posted

3. Secondary Outcome: Side Effects
Description: Evaluation of side effects
Time Frame: 6 month
Reporting Status: Not Posted

4. Secondary Outcome: Mobilisation
Description: Evaluation of time to post surgical mobilization
Time Frame: 6 month
Reporting Status: Not Posted

5. Secondary Outcome: Costs
Description: Evaluation costs between groups
Time Frame: 6 month
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Oxycodon | Patient Controlled Device With Pritramid
Serious Adverse Events (participants affected / at risk) | 0/113 | 0/126
Other Adverse Events (participants affected / at risk) | 0/113 | 0/126

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes